CLINICAL TRIAL: NCT05595057
Title: Coping, Perceived Meaning, Joy, Horizontal Civility At Work
Status: Withdrawn | Type: Observational
Why Stopped: PI no longer at institution
Sponsor: Methodist Health System (Other)
Responsible Party: Sponsor
Other Study IDs: 069.NUR.2021.A
Record Dates: First submitted 2022-02-03; First posted 2022-10-26 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2023-08

CONDITIONS: Workplace Incivility; Joy; Self Efficacy
MeSH Terms: conditions — Incivility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of this study is to assess and describe employee characteristics associated with perceived horizontal inter-collegial workplace uncivil behavior within nursing services, and identify any relationships with meaning and joy in work (MJW), and assess job satisfaction.

DETAILED DESCRIPTION:
Workplace incivility in the nursing profession interferes with the establishment of a culture of safety, places patient safety at risk, and erodes job satisfaction and a positive staff environment (Kile, Eaton, deValpine, & Gilbert, 2019). Contemporary research among nurses in Magnet and Pathway to Excellence-designated hospitals reflects that 'nurse coworker incivility is sporadic on average but varies considerably across nurses (Smith, Morin, & Lake, 2018). However, there needs to be more administrative focus and attention on nurses' work environments to support civil workplaces where the nurses focuses on and provide patient care (Smith et al., 2018). Hence, the proposed study aims to examine intra-organizational incivility, that is incivility 'originating from within the organization' (Cortina, Magley, Williams, & Langhout, 2001), and will examine nurses' intrapersonal resourcefulness to support or promote proactive self-management in a self-efficacious manner, thus ameliorating workplace incivility, dissatisfaction, and detrimental outcomes. For this study, nursing staff will include registered nurses and other para-professionals employed under nursing services. The para-professionals employed under nursing services are Mental Health Technicians (MHT), Patient Care Technicians (PCT), Surgical Technicians (ST), and Emergency Medical Services (EMS).

ELIGIBILITY:
Inclusion Criteria:

* The sample of participants will include all willing individuals who are registered nurses (full time, part time, and per-diem) or nursing para-professionals employed by MHS and working at the MDMC, MCMC, MLMC, or MMMC campuses.
* Provide direct patient care for more than 50% of work hours.
* All participants must be able to read and understand English.

Exclusion Criteria:

* Excluded from the study will be employees who do not provide direct patient care for at least 50% of the time, educators, managers, leaders, advanced practice nurses, and non-nursing service personnel.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: A power analysis using the G*Power 3.1 [1] indicated that a total sample of 84 people would be needed to detect a medium effect (Cohen's ρ= 0.30) with 80% power using exact correlation-difference from constant (one sample case) with alpha at 0.05. We plan to enroll 105 people to account for the 20% attrition rate (Faul, Erdfelder, Buchner, & Lang, 2009). Participants will be asked to respond online to a questionnaire launched via Survey Monkey® and provide demographic information and information related to coping, perceived meaning, joy, and horizontal civility at work.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2023-08-24 (Actual); Study Completion 2023-08-24 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | Dec 2021 - Dec 2022
  Self-efficacy is directly related to job satisfaction
Perceived self-efficacy | Dec 2021 - Dec 2022
  Perceived self-efficacy is inversely related to incivility
MJW | Dec 2021 - Dec 2022
  MJW is inversely related to perceived incivility [Rutledge et al, 2018]
Nursing staff in high-stress levels clinical areas and high sense of urgency (e.g., critical care and the emergency department (ED)) | Dec 2021 - Dec 2022
  Nursing staff in high-stress levels clinical areas and high sense of urgency (e.g., critical care and the emergency department (ED)) are more likely to be exposed to incivility
Years of experience in this hospital predicts staff's perception of incivility | Dec 2021 - Dec 2022
  Years of experience in this hospital predicts staff's perception of incivility
Years of experience in nursing services at any facility predicts report of coping self-efficacy | Dec 2021 - Dec 2022
  Years of experience in nursing services at any facility predicts report of coping self-efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Gret Friedrich-Cuntz, EdD, Principal Investigator — Methodist Charlton Medical Center; Cheyenne Ruby, MSN, Principal Investigator — The Methodist Hospital Research Institute; Laura Sweatt, MSN, Principal Investigator — Methodist Mansfield Medical Center; Julie Vinson, BSN, Principal Investigator — Methodist Midlothian Medical Center
Locations (4):
- United States (4):
  - Methodist Dallas Medical Center, Dallas, Texas
  - Methodist Mansfield Medical Center, Dallas, Texas
  - Methodist Charlton Family Medicine, Dallas, Texas
  - Methodist Midlothian Medical Center, Midlothian, Texas